CLINICAL TRIAL: NCT07105371
Title: Patients With ALS and Other Motor Discorders Will be Treated With Mesenchymal Cell Exosome Solution
Brief Title: Patients With ALS and Other Motor Disorders Will be Treated With Mesenchymal Cell Exosome Solution
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The Foundation for Orthopaedics and Regenerative Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FOREM2024EX01
Record Dates: First submitted 2025-07-22; First posted 2025-08-05 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Motor Disorders
Keywords: exosomes; secretome; ALS; Kennedy disease; Congenital Myasthenic Syndrome; Lewy body dementia
MeSH Terms: conditions — Motor Disorders; Bulbo-Spinal Atrophy, X-Linked; Myasthenic Syndromes, Congenital; Lewy Body Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Group (AlloEx) (Experimental)
  Interventions: Biological: AlloEx exosomes

INTERVENTIONS:
Biological: AlloEx exosomes — This is an intranasal treatment of exosomes derived from mesenchymal stem cells.

SUMMARY:
Patients with ALS and other Motor Discorders will be treated with mesenchymal cell exosome solution.

DETAILED DESCRIPTION:
Single Arm non-controlled study. Patients are prospectively evaluated then treated. Outcomes are tracked after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients will need a diagnosis established by a neurologist. Patients must be able to provide informed consent, or have a guardian who does. They must be able to travel to the site of treatment.

Exclusion Criteria:

* Patients were excluded from the trial if they were pregnant or had active cancer at the screening consultation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2024-07-14 (Actual); Primary Completion 2025-03-14 (Actual); Study Completion 2025-03-14 (Actual)

PRIMARY OUTCOMES:
ALSFRS-R Results | from enrollment until 6 months after treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Medical Surgical Associates Center, St John's, Antigua and Barbuda

REFERENCES:
- [Derived] Prodromos CC, Del Villar R, Jin MY, Abd-Elsayed A, Candido K. Exosome-rich mesenchymal stem cell secretome improves strength in patients with amyotrophic lateral sclerosis, Kennedy disease, congenital myasthenic syndrome and Lewy body dementia. Am J Stem Cells. 2025 Oct 15;14(4):217-229. doi: 10.62347/FTXA8845. eCollection 2025. PMID 41278139